CLINICAL TRIAL: NCT04892888
Title: Special Use Results Survey: Spikevax Intramuscular Injection (Previously COVID-19 Vaccine Moderna Intramuscular Injection) for Subjects With Underlying Disease Considered to be at High Risk for Severe Illness, Acute Phase Safety Surveillance (COVID-19)
Brief Title: Survey of the Moderna COVID-19 Vaccine in People at High-Risk of Developing Severe COVID-19 Symptoms
Status: Withdrawn | Type: Observational
Why Stopped: Business decision
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: PNR-1475; jRCT2031210095 (Registry Identifier: jRCT)
Record Dates: First submitted 2021-05-18; First posted 2021-05-19 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Coronavirus Disease (COVID-19)
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 Vaccine Intramuscular Injection 0.5 mL: COVID-19 vaccine intramuscular injection, 2 doses of 0.5 mL per dose administered intramuscularly at an interval of 4 weeks.
  Interventions: Biological: COVID-19 Vaccine

INTERVENTIONS:
Biological: COVID-19 Vaccine — COVID-19 Vaccine Intramuscular Injection
  Other Names: COVID-19 Vaccine Moderna Intramuscular Injection; Spikevax Intramuscular Injection

SUMMARY:
This study is a survey of the Moderna COVID-19 vaccine in Japanese people at high risk of developing severe COVID-19 symptoms. The study sponsor will not be involved in how the participants are treated but will provide instructions on how the clinics will record what happens during the study.

The main aim of the study is to check for side effects of the Moderna COVID-19 vaccine in this group. This will be from the first vaccination to 28 days after the second vaccination.

The number of visits to the clinic will depend on the clinic's standard practice.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is capable of understanding the contents of the investigation, recording his/her own symptoms in the health observation diary, and has obtained written consent to participate in the investigation from the vaccinee himself/herself (If minor, parent or legal guardian).
2. The participant has an underlying disease at the time of this drug vaccination that is considered to pose a high risk of aggravation of COVID-19.

Exclusion Criteria:

1. The subject has any contraindication to this drug.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population of this survey are vaccinees who meet the inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with at least One Adverse Events (AEs) | 56 days
  An adverse event (Adverse Event: AE) is any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product. It does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (Including laboratory abnormalities), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Percentage of Participants with Specified AEs (Local Reactions) at the Vaccination Site | 56 days
  Specified AEs (Local reactions) at the vaccination site are defined as injection site pain, redness and swelling. The participants will evaluate the symptoms at the vaccination site (local reactions) and systemic symptoms (systemic events) and will record with the health observation diary. Percentage of participants with specified AEs (local reactions) at the vaccination site will be reported.
Percentage of Participants with Specified AEs (Systemic Events) | 56 days
  Specified AEs (Systemic events) are defined as vomiting, diarrhoea, headache, malaise, chills, myalgia, and arthralgia. The participants will evaluate the symptoms at the vaccination site (local reactions) and systemic symptoms (systemic events) and will record with the health observation diary. Percentage of participants with specified AEs (systemic events) at the vaccination site will be reported.

SECONDARY OUTCOMES:
Number of Participants who Take COVID-19 Pathogen (SARS-COV-2) Test during the Study | 56 days
Number of Participants who Developed COVID-19 during the Study | 56 days
Number of Participants Who Have Sever COVID-19 Infection during the Study Evaluated by Investigator | 56 days
  Number of participants who have sever COVID-19 infection during the study evaluated by investigator will be reported. Investigator will evaluate the severity of COVID-19 infection with COVID-19 information entered in the case report form in reference to "Guidance for Clinical Practice of Novel Coronavirus Infection (COVID-19)".

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Takeda Selected Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/61443d95c15195002c0ba2ee?idFilter=%5B%22PNR-1475%22%5D